CLINICAL TRIAL: NCT04148716
Title: Identification and Characterization of microRNAs Involved in Esophageal, Gastric and Duodenal Fibrotic Manifestations of Systemic Scleroderma
Brief Title: microRNAs in Systemic Scleroderma
Acronym: Dig-ScS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 19-AOI-07
Record Dates: First submitted 2019-10-25; First posted 2019-11-01 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: recruitement of 9 patients
  Interventions: Procedure: additional biopsies
- control: recruitement of 9 control person
  Interventions: Procedure: additional biopsies

INTERVENTIONS:
Procedure: additional biopsies — additional biopsies during a fibroscopy planned in the care

SUMMARY:
No studies have investigated the expression of miRNAs in Dig-ScS tissues. In the absence of specific treatment for this frequent impairment in this connectivity, the team proposes to study miRNA profiles in the esophagus and duodenum to identify new therapeutic targets. The team is studying the involvement of pro-fibrotic "key" miRNAs called "FibromiRs", including 3 miRNAs from the DNM3os locus (miR-199a-3p, miR-199a-5p and miR-214 - characterized by the host laboratory) associated with monitoring the response to TGF-β in fibroblasts and their potential interaction with pharmacological treatments such as nintedanib and/or PPARγ agonists. The approach is part of a pilot study that can lead to a larger project after validation of the hypotheses.

It also seems interesting to make a precise anatomopathological description with a gradation of the digestive fibrotic damage in view of the paucity of medical literature in this field

ELIGIBILITY:
Patient Inclusion Criteria

* Subject aged between 18 and 75 years old, meeting the 2013 ACR/EULAR classification criteria for ScS
* Subject under an indication for the performance of esogastro-duodenal fibroscopy (FOGD), the main ones being: anemia, anorexia, weight loss, gastroesophageal reflux disease, dysphagia or odynophagia, ulcer syndrome, suspected portal hypertension
* Supported at Nice University Hospital
* Subject understands and speaks French and is able to give written consent
* Subject affiliated to Social Security or a similar scheme
* Subjects accepting additional digestive biopsies

Control inclusion criteria:

* Subject aged between 18 and 75 years old, without dysimmunitary disease
* Subject within the scope of an indication for the performance of a FOGD as defined by the treating gastroenterologist
* Subject accepting to be serologically tested for HIV and HCV
* Subject understands and speaks French and is able to give written consent
* Subject affiliated to Social Security or a similar scheme
* Subjects accepting additional digestive biopsies

Exclusion Criteria:

* Subject protected by law under guardianship or curatorship, or unable to participate in a clinical study under Article L. 1121-16 of the French Public Health Code
* Subject who has participated in a clinical research study in the last 3 months in which he/she was exposed to a pharmaceutical product or medical device
* Subject who has stayed in a tropical or subtropical country in the last 3 months
* Pregnant or breastfeeding participant
* Subject on a special diet for medical reasons and prescribed by a doctor or dietician (e.g. a low-calorie diet or a diet designed to lower cholesterol levels)
* Subject who regularly consumes large quantities of alcohol, i. e. more than 50 g of pure alcohol per day (e. g. more than 4 glasses of 150 ml wine, more than 4 pints of 250 ml beer, or more than 4 glasses of 40 ml containing strong alcohol)
* Subject who has used an illegal recreational drug in the past 3 months
* Subject who has taken an immunosuppressive or immunomodulatory drug (excluding corticosteroids administered at doses ≤ 10 mg/d PREDNISONE equivalent) within the previous 2 weeks, or for more than 14 consecutive days within the last 3 months
* Subject who has been vaccinated within the last 3 months
* Subject who received a blood transfusion or immunoglobulins in the last 3 months
* Subject stating that he has not been fasting for at least 10 hours
* Subject reporting HIV or HCV status
* Subject who had an infectious episode or was treated with antibiotics during the 4 weeks prior to the visit
* Subject with a positive pregnancy test
* Subject with graft versus host disease, or who has received therapy involving hematopoietic stem cells
* Subject with a severe and/or chronic and/or recurrent pathology, in particular:
* A chronic inflammatory disease of the intestine (Crohn's disease, ulcerative colitis), epidermis (psoriasis, atopic dermatitis), joints (rheumatoid arthritis), nervous system (multiple sclerosis); except ScS.
* A neurodegenerative disease
* Diabetes mellitus
* Subject who has been diagnosed with cancer and has not been in remission for more than 5 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people needed esogastro-duodenal fibroscopy
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
description of the profile of miR based expression on cytokinic treatments and stimuli. | 4 years
  fundamental research aimed at determining an expression profile of miR as a function of cytokinic treatments and stimuli. proteins (cytokins) study to describe the profil of miR

CONTACTS AND LOCATIONS:
Locations (1):
- Nice Hospital, Nice, France